CLINICAL TRIAL: NCT01499199
Title: A Single-arm Study of the Safety, Efficacy and Central Nervous System and Plasma PK of GSK1349572 (Dolutegravir, DTG) 50 mg Once Daily in Combination With the Abacavir/Lamivudine Fixed Dose Combination Tablet Over 96 Weeks in HIV-1 Infected Antiretroviral Naive Adult Subjects
Brief Title: A Study of the Pharmacokinetics and Antiviral Activity of Dolutegravir in the Central Nervous System in HIV-1 Infected ART-naive Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116070
Record Dates: First submitted 2011-12-15; First posted 2011-12-26 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-01

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: cerebrospinal fluid (CSF); ART-naive; integrase inhibitor; dolutegravir; antiretroviral therapy naive
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dolutegravir 50mg Once Daily (Experimental): All subjects will receive 50mg dolutegravir once daily in combination with background antiretroviral therapy consisting of one abacavir/lamivudine fixed dose combination tablet once daily
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — 50mg Once Daily

SUMMARY:
ING116070 is a Phase IIIb single-arm, open-label, multicenter study. The study will be conducted in approximately 14 HIV-1 infected antiretroviral therapy (ART)-naïve subjects. Subjects who fulfill eligibility requirements will receive dolutegravir (DTG) 50 mg once daily in combination with the fixed dose dual nucleoside reverse transcripatase inhibitor(NRTI) abacavir/lamivudine (ABC/3TC) for 96 weeks. One pair of pharmacokinetic (PK) samples in plasma and cerebral spinal fluid (CSF) (matching time) for determination of DTG concentration will be collected at Week 2 and Week 16. Samples for plasma HIV-1 RNA will be collected at Baseline and various time points throughout the study and samples for HIV-1 RNA levels in the CSF will be collected at Baseline, Week 2 and Week 16. Safety, additional measures of antiviral activity and development of viral resistance will also be evlauated. The primary analysis will take place after the last subject completes 16 weeks on therapy; additional analyses will be conducted after the last subject completes Weeks 2 and 96 (end of study).

DETAILED DESCRIPTION:
ING116070 is a Phase IIIb single-arm, open-label, multicenter study. The study will be conducted in approximately 14 HIV-1 infected antiretroviral therapy (ART)-naïve subjects. Subjects who meet all screening requirements may enter the study and initiate treatment as soon as all screening procedures have been completed and results are available and on file. The 14-day screening period may be extended to 28 days to allow receipt of all Screening assessment results and to accommodate scheduling.

Subjects who fulfill eligibility requirements will receive dolutegravir (DTG) 50 mg once daily in combination with the fixed dose dual nucleoside reverse transcripatase inhibitor(NRTI) abacavir/lamivudine ABC/3TC for 96 weeks. One pair of pharmacokinetic (PK) samples in plasma and CSF (matching time) for determination of DTG concentration will be collected at Week 2 and Week 16. Samples for plasma HIV-1 RNA will be collected at Baseline and various time points throughout the study and samples for HIV-1 RNA levels in the CSF will be collected at Baseline, Week 2 and Week 16. Safety, additional measures of antiviral activity and development of viral resistance will also be evlauated. The primary analysis will take place after the last subject completes 16 weeks on therapy; additional analyses will be conducted after the last subject completes Weeks 2 and 96 (end of study).

Subjects are considered to have completed the study if they remain on therapy (i.e., have not permanently discontinued investigational product [IP]) and complete the Treatment Phase, including the Week 96 visit.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults at least 18 years of age. Females are eligible to enter and participate in the study if she is (1) of non-childbearing potential or (2) of childbearing potential with a negative pregnancy test at Screening and Day 1 and agrees to use protocol-defined methods of birthcontrol while on the study.
* HIV-1 infection as documented by Screening plasma HIV-1 RNA greater than or equal to 5000 copies/mL
* CD4+ cell count greater than or equal to 200 cells/mm3
* Antiretroviral-naive (less than or equal to 10 days of prior therapy with any antiretroviral agent following diagnosis of HIV-1 infection)
* Signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening
* Documentation that the subject has been screened for, and is negative for the HLA-B*5701 allele
* Is willing to undergo serial lumbar punctures

Exclusion Criteria:

* Relative or absolute contraindication to lumbar puncture, such as current coagulopathy, thrombocytopenia (platelets less than 50,000/microliter), hemophilia, or use of anticoagulant medication
* Moderate or severe cognitive impairment
* Women who are pregnant or breastfeeding
* Any evidence of an active Center for Disease Control and Prevention (CDC) Category C disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy or historic CD4+ cell levels less than 200cells/mm3
* Subjects with any degree of hepatic impairment
* Positive for Hepatitis B at screening (+HbsAg), or an anticipated need for Hepatitis C virus (HCV) therapy during the study
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the subject
* Recent history (less than or equal to 3 months) of any upper or lower gastrointestinal bleed, with the exception of anal or rectal bleeding
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with any of the following agents within 28 days of Screening: radiation therapy, cytotoxic chemotherapeutic agents, any immunomodulators that alter immune responses
* Treatment with any agent, except recognized ART as allowed above, with documented activity against HIV-1 in vitro within 28 days of first dose of IP
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of IP
* Any evidence of primary viral resistance based on the presence of any major resistance-associated mutation in the Screening result or, if known, any historical resistance test result. Note: retests of Screening genotypes are not allowed
* Any verified Grade 4 laboratory abnormality (a single repeat test is allowed during the Screening period to verify a result). Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound is exclusionary
* Alanine aminotransferase (ALT) greater than 5 times the upper limit of normal (ULN)
* ALT greater than or equal to 3xULN and bilirubin greater than or equal to 1.5xULN (with greater than 35% direct bilirubin)
* Subject has creatinine clearance of less than 50 mL/min via Cockroft-Gault method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (3):
- United States (3):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Providence, Rhode Island

REFERENCES:
- [Background] Letendre S, Mills A, Tashima K, et al. Distribution and antiviral activity in cerebrospinal fluid (CSF) of the integrase inhibitor, dolutegravir (DTG): ING116070 week 16 results. Published at: Conference on Retroviruses and Opportunistic Infections - 20th Annual; March 3-6, 2013; Atlanta, GA.
- [Background] Letendre S, Mills A, Tashima K, et al. CSF penetration and antiviral activity of the integrase inhibitor, dolutegravir (DTG, GSK1349572): ING116070 week 16 results. Published at: International Symposium on Neuropsychiatry & HIV - 6th; May 9-10, 2013; Barcelona, Spain
- [Derived] Letendre SL, Mills AM, Tashima KT, Thomas DA, Min SS, Chen S, Song IH, Piscitelli SC; extended ING116070 study team. ING116070: a study of the pharmacokinetics and antiviral activity of dolutegravir in cerebrospinal fluid in HIV-1-infected, antiretroviral therapy-naive subjects. Clin Infect Dis. 2014 Oct;59(7):1032-7. doi: 10.1093/cid/ciu477. Epub 2014 Jun 18. PMID 24944232

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants received dolutegravir (DTG ) 50 milligrams (mg) once daily (OD) in combination with abacavir/lamivudine (ABC/3TC) for 96 weeks.
Groups:
- Dolutegravir 50 mg OD: Participants received dolutegravir (DTG) 50 milligrams (mg) once daily (OD) in combination with abacavir/lamivudine (ABC/3TC) OD.
Period: Overall Study
Arm/Group | Dolutegravir 50 mg OD
Started | 13
Completed | 11
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (6.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13
Baseline plasma human immunodeficiency virus-1 (HIV-1) ribonucleic acid (RNA) [Median (Full Range); unit: log10 copies/mL] — The absolute value of plasma HIV-1 RNA was measured at Baseline as log10 copies/milliliter (mL).
  log10 copies/mL | 4.73 [3.60 to 6.57]
Number of participants with Baseline plasma HIV-1 RNA <=100000 copies/mL and >100000 copies/mL [Number; unit: Participants] — The number of participants with Baseline plasma HIV-1 RNA <= 100000 copies/mL and >100000 copies/mL was measured.
  Participants
    <=100000 copies/mL | 8
    >100000 copies/mL | 5

OUTCOME MEASURES:

1. Primary Outcome: The Ratio of Total and Unbound DTG Concentrations Between Cerebrospinal Fluid (CSF) and Plasma at Week 2 and Week 16
Description: Cerebrospinal fluid (CSF) is a clear, colorless bodily fluid produced in the choroid plexus of the brain. The CFS samples were collected at the Week 2 and Week 16 visits, within 1 hour of plasma pharmacokinetic (PK) sampling. The ratio (presented as a percentage) of CSF DTG concentration over paired plasma total DTG concentration (RCSF_plasma) was calculated at the Week 2 and Week 16 visits.
Time Frame: Week 2 and Week 16
Population: Plasma/CSF DTG Paired Sample Population: participants (par.) with plasma and CSF samples collected post-dose and within 1 hour of each other (one par. withdrew prior to Week 2 and did not contribute to PK assessments). One par. was excluded from the analysis at Week 2 because his/her paired samples were not collected within the specified timeframe.
Measure: Median (Full Range); unit: percentage
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 12
percentage
  Week 2, n=11 | 0.516 [0.115 to 0.658]
  Week 16, n=12 | 0.412 [0.299 to 2.04]

2. Primary Outcome: Total DTG Plasma Concentrations at Week 2 and Week 16
Description: Total plasma DTG concentrations were calculated at the Week 2 and Week 16 visits.
Time Frame: Week 2 and Week 16
Population: Plasma DTG Concentration Population: all participants receiving DTG who underwent PK sampling during the study and provided evaluable DTG plasma concentration data
Measure: Median (Full Range); unit: Micrograms per milliliter (µg/mL)
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 12
Micrograms per milliliter (µg/mL)
  Week 2 | 3.36 [2.09 to 5.28]
  Week 16 | 3.21 [0.64 to 4.92]

3. Primary Outcome: Unbound DTG Plasma Concentrations at Week 2 and Week 16
Description: Unbound (free, not bound to cellular proteins) plasma DTG concentrations were calculated at the Week 2 and Week 16 visits.
Time Frame: Week 2 and Week 16
Population: Plasma DTG Concentration Population
Measure: Median (Full Range); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 12
Nanograms per milliliter (ng/mL)
  Week 2 | 17.1 [10.3 to 24.0]
  Week 16 | 23.9 [3.81 to 32.1]

4. Primary Outcome: Plasma DTG Unbound Fraction at Week 2 and Week 16
Description: The unbound fraction of DTG in plasma (presented as a percentage of unbound [i.e., free DTG not bound to cellular proteins] DTG plasma concentration over paired plasma total DTG concentration) was calculated at the Week 2 and Week 16 visits.
Time Frame: Week 2 and Week 16
Population: Plasma DTG Concentration Population
Measure: Median (Full Range); unit: Percentage
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 12
Percentage
  Week 2 | 0.488 [0.333 to 0.655]
  Week 16 | 0.701 [0.488 to 4.30]

5. Primary Outcome: DTG Concentrations in CSF at Weeks 2 and Week 16
Description: CSF is a clear, colorless bodily fluid produced in the choroid plexus of the brain. The CFS samples were collected at the Week 2 and Week 16 visits, within 1 hour of plasma PK sampling. DTG concentration in CSF were calculated at the Week 2 and Week 16 visits.
Time Frame: Week 2 and Week 16
Population: CSF DTG Concentration Population: all participants receiving DTG who underwent lumbar puncture during the study and provided evaluable DTG CSF concentration data. One participant was excluded from the analysis at Week 2.
Measure: Median (Full Range); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 12
Nanograms per milliliter (ng/mL)
  Week 2, n=11 | 18.2 [4.0 to 23.2]
  Week 16, n=12 | 13.2 [3.7 to 18.3]

6. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <50 Copies Per Milliliter (c/mL) at Baseline and Weeks 2, 4, 8, 12, and 16
Description: HIV-1 RNA response in plasma was measured as the number of participants with HIV-1 RNA less than 50 c/mL at Baseline, Week 2, Week 4, Week 8, Week 12, and Week 16.
Time Frame: Baseline; Weeks 2, 4, 8, 12, and 16
Population: Intent -to-Treat Exposed (ITT-E) Population: all participants who received at least one dose of investigational product
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
participants
  Baseline | 0
  Week 2 | 4
  Week 4 | 6
  Week 8 | 8
  Week 12 | 10
  Week 16 | 10

7. Secondary Outcome: Absolute Values and Change From Baseline in Plasma Human Immunodeficiency Virus (HIV-1) Ribonucleic Acid (RNA) Levels at Weeks 2, 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, and 96
Description: The plasma samples were collected at the Week 2, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, and Week 96 visits. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 2, 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, and 96
Population: ITT-E Population. Only those participants available at the indicated time point were assessed.
Measure: Median (Full Range); unit: log10 copies/mL
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
log10 copies/mL
  Absolute value, Baseline, n=13 | 4.73 [3.60 to 6.57]
  Absolute value, Week 2, n=12 | 2.05 [1.59 to 2.99]
  Change from Baseline, Week 2, n=12 | -2.53 [-3.70 to -2.01]
  Absolute value, Week 4, n=12 | 1.67 [1.59 to 2.49]
  Change from Baseline, Week 4, n=12 | -3.04 [-4.08 to -2.01]
  Absolute Value, Week 8, n=12 | 1.59 [1.59 to 2.48]
  Change from Baseline, Week 8, n=12 | -3.10 [-4.09 to -2.01]
  Absolute value, Week 12, n=12 | 1.59 [1.59 to 2.36]
  Change from Baseline, Week 12, n=12 | -3.04 [-4.20 to -2.01]
  Absolute value, Week 16, n=12 | 1.59 [1.59 to 2.37]
  Change from Baseline, Week 16, n=12 | -3.04 [-4.19 to -2.01]
  Absolute Value, Week 24, n=12 | 1.59 [1.59 to 2.21]
  Change from Baseline, Week 24, n=12 | -3.11 [-4.35 to -2.01]
  Absolute value, Week 36, n=11 | 1.59 [1.59 to 1.62]
  Change from Baseline, Week 36, n=11 | -3.08 [-3.89 to -2.01]
  Absolute value, Week 48, n=11 | 1.59 [1.59 to 2.10]
  Change from Baseline, Week 48, n=11 | -3.00 [-3.78 to -2.01]
  Absolute value, Week 60, n=11 | 1.59 [1.59 to 2.19]
  Change from Baseline, Week 60, n=11 | -3.00 [-3.89 to -2.01]
  Absolute value, Week 72, n=11 | 1.59 [1.59 to 2.01]
  Change from Baseline, Week 72, n=11 | -3.08 [-3.78 to -2.01]
  Absolute value, Week 84, n=11 | 1.59 [1.59 to 1.72]
  Change from Baseline, Week 84, n=11 | -3.08 [-3.89 to -1.88]
  Absolute value, Week 96, n=11 | 1.59 [1.59 to 3.05]
  Change from Baseline, Week 96, n=11 | -3.08 [-3.78 to -0.55]

8. Secondary Outcome: Number of Participants With CSF HIV-1 RNA <50 Copies/Milliliter (c/mL) at Baseline, Week 2, and Week 16
Description: The antiviral activity of dolutegravir in CSF over time was measured as the number of participants with HIV-1 RNA <50 copies/milliliter (c/mL).
Time Frame: Baseline, Week 2, and Week 16
Population: CSF Pharmacodynamic Population: all participants who received DTG and underwent lumbar puncture during the study and provided CSF HIV-1 RNA data. Only those participants available at the indicated time points were assessed.
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
participants
  Baseline, n=13 | 1
  Week 2, n=12 | 7
  Week 16, n=11 | 11

9. Secondary Outcome: Absolute Values and Change From Baseline in CSF HIV-1 RNA Levels at Week 2 and Week 16
Description: The antiviral activity of dolutegravir in CSF over time was measured as absolute values and change from Baseline in HIV-1 RNA levels in CSF at Week 2 and Week 16. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline, Week 2, and Week 16
Population: CSF Pharmacodynamic Population. Only those participants available at the indicated time points were assessed.
Measure: Median (Full Range); unit: log10 c/mL
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
log10 c/mL
  Absolute value, Baseline, n=13 | 3.64 [1.46 to 5.60]
  Absolute value, Week 2, n=12 | 0.98 [0.00 to 3.30]
  Change from Baseline, Week 2, n=12 | -2.19 [-3.11 to -1.29]
  Absolute value, Week 16, n=11 | 0.00 [0.00 to 0.70]
  Change from Baseline, Week 16, n=11 | -3.42 [-5.60 to -1.46]

10. Secondary Outcome: Number of Participants With the Indicated Number of Copies of HIV-1 RNA in Both the CSF and Plasma at Baseline, Week 2, and Week 16
Description: The relationship between HIV-1 RNA suppression in plasma and the CSF was measured as a comparison and as a change in the number of participants in the cross tabulation of <50 copies/mL in plasma, <50 copies/mL in CSF, >=50 copies/mL in plasma, and >=50 copies/mL in CSF at Baseline, Week 2, and Week 16.
Time Frame: Baseline, Week 2, and Week 16
Population: CSF Pharmacodynamic Population. Only those participants available at the indicated time point were assessed.
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
participants
  Baseline, CSF<50 c/mL, Plasma<50 c/mL, n=13 | 0
  Baseline, CSF<50 c/mL, Plasma>=50 c/mL, n=13 | 1
  Baseline, CSF>=50 c/mL, Plasma<50 c/mL, n=13 | 0
  Baseline, CSF>=50 c/mL, Plasma>=50 c/mL, n=13 | 12
  Week 2, CSF<50 c/mL, Plasma<50 c/mL, n=12 | 4
  Week 2, CSF<50 c/mL, Plasma>=50 c/mL, n=12 | 3
  Week 2, CSF>=50 c/mL, Plasma<50 c/mL, n=12 | 0
  Week 2, CSF>=50 c/mL, Plasma>=50 c/mL, n=12 | 5
  Week 16, CSF<50 c/mL, Plasma<50 c/mL, n=11 | 9
  Week 16, CSF<50 c/mL, Plasma>=50 c/mL, n=11 | 2
  Week 16, CSF>=50 c/mL, Plasma<50 c/mL, n=11 | 0
  Week 16, CSF>=50 c/mL, Plasma>=50 c/mL, n=11 | 0

11. Secondary Outcome: Pearson Correlation Between CSF DTG Concentration and Absolute Values and Change From Baseline (CFB) in CSF HIV-1 RNA at Week 2, Week 16, and Overall
Description: The Pearson Correlation Coefficient is a measure of the correlation between CSF DTG concentrations and absolute values/changes from Baseline in CSF HIV-1 RNA at Week 2 and Week 16. CSF HIV-1 RNA is measured as log10 copies per milliliter (copies/mL).
Time Frame: From Baseline to Week 16
Population: CSF Pharmacodynamic Population. The overall analysis combines Week 2 and Week 16 data; thus, analysis was performed on 22 data points from 11 participants.
Measure: Mean (90% Confidence Interval); unit: Pearson Correlation Coefficient
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 11
Pearson Correlation Coefficient
  Week 2, Absolute Log10 CSF HIV-1 RNA, n=11 | 0.567 [0.062 to 0.841]
  Week 2, CFB Log10 CSF HIV-1, n=11 | 0.007 [-0.518 to 0.529]
  Week 16, Absolute Log10 CSF HIV-1 RNA, n=11 | -0.775 [-0.924 to -0.423]
  Week 16, CFB Log10 CSF HIV-1, n=11 | -0.354 [-0.740 to 0.209]
  Overall, Absolute Log10 CSF HIV-1 RNA, n=11 | 0.517 [0.193 to 0.740]
  Overall, CFB Log10 CSF HIV-1, n=11 | 0.106 [-0.265 to 0.449]

12. Secondary Outcome: Absolute Values and Change From Baseline in Cluster of Differentiation 4+ (CD4+) Cell Counts at Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, and 96
Description: The absolute value for CD4+ cell count (cells per millimeters cubed [mm^3]) was assessed at Baseline, Week 4, Week 8, Week 12, Week 16, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, and Week 96. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84, and 96
Population: ITT-E Population. Only those participants available at the indicated time point were assessed.
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
cells/mm^3
  Absolute CD4+ cell count, Baseline, n=13 | 260 [152 to 863]
  Absolute CD4+ cell count, Week 4, n=12 | 578 [374 to 903]
  Absolute CD4+ cell count, Week 8, n=12 | 645 [364 to 1118]
  Absolute CD4+ cell count, Week 12, n=12 | 589 [303 to 1144]
  Absolute CD4+ cell count, Week 16, n=12 | 573 [436 to 1156]
  Absolute CD4+ cell count, Week 24, n=12 | 634 [448 to 1339]
  Absolute CD4+ cell count, Week (Wk) 36, n=11 | 706 [534 to 1351]
  Absolute CD4+ cell count, Week 48, n=11 | 666 [537 to 939]
  Absolute CD4+ cell count, Week 60, n=11 | 702 [567 to 1266]
  Absolute CD4+ cell count, Week 72, n=11 | 823 [620 to 1315]
  Absolute CD4+ cell count, Week 84, n=11 | 907 [512 to 1341]
  Absolute CD4+ cell count, Week 96, n=11 | 843 [339 to 1436]
  Change from Baseline CD4+ cell count, Week 4, n=12 | 162 [-158 to 365]
  Change from Baseline CD4+ cell count, Week 8, n=12 | 247 [44 to 551]
  Change from Baseline CD4+ cell count, Wk 12, n=12 | 263 [-17 to 500]
  Change from Baseline CD4+ cell count, Wk 16, n=12 | 226 [-248 to 629]
  Change from Baseline CD4+ cell count, Wk 24, n=12 | 264 [86 to 762]
  Change from Baseline CD4+ cell count, Wk 36, n=11 | 480 [174 to 774]
  Change from Baseline CD4+ cell count, Wk 48, n=11 | 311 [-80 to 541]
  Change from Baseline CD4+ cell count, Wk 60, n=11 | 382 [5 to 708]
  Change from Baseline CD4+ cell count, Wk 72, n=11 | 519 [260 to 651]
  Change from Baseline CD4+ cell count, Wk 84, n=11 | 543 [94 to 792]
  Change from Baseline CD4+ cell count, Wk 96, n=11 | 467 [-65 to 859]

13. Secondary Outcome: Absolute Values and Change From Baseline in Cluster of Differentiation 8+ (CD8+) Cell Counts at Weeks 4, 12, 16, 24, 48, and 96
Description: The absolute value for CD48+ cell count (cells per millimeters cubed [mm^3]) was assessed at Baseline, Week 4, Week 12, Week 16, Week 24, Week 48, and Week 96. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 4, 12, 16, 24, 48, and 96
Population: ITT-E Population. Only those participants available at the indicated time point were assessed.
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
cells/mm^3
  Absolute CD8+ cell count, Baseline, n=13 | 757 [276 to 2945]
  Absolute CD8+ cell count, Week 4, n=12 | 874 [542 to 1984]
  Absolute CD8+ cell count, Week 12, n=12 | 865 [419 to 1472]
  Absolute CD8+ cell count, Week 16, n=12 | 706 [478 to 1818]
  Absolute CD8+ cell count, Week 24, n=11 | 876 [434 to 1634]
  Absolute CD8+ cell count, Week 48, n=11 | 708 [530 to 1318]
  Absolute CD8+ cell count, Week 96, n=11 | 842 [249 to 1582]
  Change from Baseline CD8+ cell count, Week 4, n=12 | 104 [-1123 to 1060]
  Change from Baseline CD8+ cell count,Week 12, n=11 | -53 [-1627 to 631]
  Change from Baseline CD8+ cell count,Week 16, n=11 | -35 [-1614 to 684]
  Change from Baseline CD8+ cell count,Week 24, n=11 | 235 [-418 to 710]
  Change from Baseline CD8+ cell count,Week 48, n=11 | 106 [-747 to 441]
  Change from Baseline CD8+ cell count,Week 96, n=11 | 85 [-424 to 677]

14. Secondary Outcome: Number of Participants With Post-Baseline HIV-1-associated Conditions, Including Recurrences
Description: The number of participants who reported a new or recurrent Centers for Disease Control and Prevention (CDC) Class B or Class C condition was assessed from Baseline though the date the last participant completed Week 96 + the follow-up visit (if applicable). Category (CAT) A: one or more of the following conditions (CON), without any CON listed in Categories B and C: asymptomatic HIV infection, persistent generalized lymphadenopathy, acute (primary) HIV infection with accompanying illness or history of acute HIV infection. CAT B: symptomatic CON that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or that are considered by physicians to have a clinical course or to require management that is complicated by HIV infection; and not included among CON listed in clinical CAT C. CAT C: the clinical CON listed in the AIDS surveillance case definition.
Time Frame: Baseline through the date the last participant completed Week 96 + follow-up visit (if applicable)
Population: ITT-E Population
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
participants
  New CDC Category B event | 0
  Recurring CDC Category B event | 0
  New CDC Category C event | 0
  Recurring CDC Category C event | 0

15. Secondary Outcome: The Numbers of Participants (Par.) With Clinical Adverse Events or Laboratory Abnormalities
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Refer to the general Adverse AE/SAE module for a complete list of AEs/SAEs. Any abnormal laboratory test result (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g., electrocardiograms [ECGs], radiological scans, vital sign measurements), including those that worsen from Baseline, and were felt to be clinically significant in the medical and scientific judgment of the investigator, were recorded as AEs or SAEs. Clinically suspected cases of hypersensitivity to ABC were also SAEs.
Time Frame: Baseline (BL) through the date the last participant completed Week (W) 96 + the follow-up visit (if applicable)
Population: Safety Population: all participants who received at least one dose of study medication. Participants were analyzed according to the actual treatments received. Participants were not excluded from this population as a result of changes to the background regimen.
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
participants
  Any AE | 13
  Clinical chemistry toxicities | 12
  Hematology toxicities | 3
  Abnormal ECG (clinically significant) | 0

16. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic and Phenotypic Resistance to DTG and Other Antiretroviral Therapy (ART)
Description: The number of participants with treatment-emergent genotypic and phenotypic resistance to integrase inhibitors (INIs), nucleoside reverse transcriptase inhibitors (NRTIs), non-nucleoside reverse transctiptase inhibitors (NNRTIs), and protease inhibitors (PIs) was assessed.
Time Frame: Baseline through the date the last participant completed Week 96
Population: Protocol Defined Virologic Failure (PDVF) Genotypic Population (Integrase inhibitor [IN] Results at Baseline and PDVF): The PDVF Genotypic and Phenotypic populations consisted of all participants in the ITT-E Population with available on-treatment genotypic and phenotypic resistance data, respectively, at the time of PDVF
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50 mg OD
Number analyzed (Participants) | 13
participants
  Treatment-emergent genotypic resistance | 0
  Treatment-emergent phenotypic resistance | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study medication to the date the last participant completed Week 96+ follow-up visit (if applicable).
Description: SAEs and non-serious AEs were reported for members of the Safety Population, comprised of all participants randomized to treatment who received at least one dose of trial medication during the treatment period.
Arm/Group | Dolutegravir 50 mg OD
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dolutegravir 50 mg OD (N=13)
Pharyngitis (Infections and infestations) | 1
Cholecystitis (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dolutegravir 50 mg OD (N=13)
Folliculitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 5
Anal chlamydia infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Otitis externa (Infections and infestations) | 1
Syphilis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Headache (Nervous system disorders) | 7
Carpal tunnel syndrome (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
Hunger (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 1
Eye pruritus (Eye disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 3
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Acarodermatitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 2
Herpes simplex (Infections and infestations) | 2
Oropharyngeal gonococcal infection (Infections and infestations) | 2
Body tinea (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Chlamydial infection (Infections and infestations) | 1
Gonorrhoea (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Sciatica (Nervous system disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Impaired healing (General disorders) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 1
Lipase increased (Investigations) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Emotional disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Urine flow decreased (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.